CLINICAL TRIAL: NCT01655810
Title: Vitamin D and Early Markers of Cardiovascular Disease in African Americans
Brief Title: Vitamin D, Cardiovascular Disease, and African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201102160
Record Dates: First submitted 2012-07-19; First posted 2012-08-02 (Estimated); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Vitamin D Deficiency; Type 2 Diabetes Mellitus; Cardiovascular Disease
MeSH Terms: conditions — Vitamin D Deficiency; Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D 4000 IU (Active Comparator): PO daily
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate
- Vitamin D 600 IU (Active Comparator): PO daily
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Multivitamin containing cholecalciferol 4000 units orally daily
  Other Names: Cholecalciferol
  Arms: Vitamin D 4000 IU
Dietary Supplement: Vitamin D3 — Multivitamin containing cholecalciferol 600 units orally daily
  Other Names: Cholecalciferol
  Arms: Vitamin D 600 IU
Dietary Supplement: Calcium carbonate — 500 mg orally twice daily

SUMMARY:
African-Americans have higher rates of cardiovascular disease morbidity and mortality, as well as vitamin D deficiency. Multiple observational studies have demonstrated an increased risk of vitamin D deficiency in African Americans with type 2 diabetes and correlation between cardiovascular disease and vitamin D levels; however, there is a lack of interventional trials exploring this connection. The objective of this proposal is to address the hypothesis that treatment of vitamin D deficiency in African Americans with type 2 diabetes will improve subclinical markers of cardiovascular disease.

DETAILED DESCRIPTION:
This study will be a double blinded, randomized controlled trial of vitamin D3 supplementation, 4,000 international units per day versus 600 international units per day, for one year to determine the effects on markers of subclinical cardiovascular disease in African Americans with type 2 diabetes and vitamin D deficiency. Outcome assessment will focus on changes in carotid intima-medial thickness (CIMT - ultrasound of the thickness of blood vessels in the neck), as well as markers of systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* African Americans of both genders
* Age 50-70 years
* Type 2 diabetes (A1C < 9.0%), on stable therapy with oral medications, insulin, or a combination
* 25(OH)D level < 20 ng/ml
* BP < 140/90 mmHg; LDL < 140 mg/dl

Exclusion Criteria:

* Pregnancy
* Cardiovascular disease
* Stage 3 or worse chronic kidney disease
* High urine or serum calcium or history of recurrent kidney stones
* Unstable medical conditions or major systemic diseases such as malignancy

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-08-13 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in carotid intima-medial thickness | 0, 6, and 12 months

SECONDARY OUTCOMES:
Change from baseline in systemic inflammatory markers | 0, 6, and 12 months
Serum calcium | 0, 1, 3, 6, 9, and 12 months
Urinary Calcium | 0, 1, 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Bernal-Mizrachi, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States